CLINICAL TRIAL: NCT02451332
Title: Prenatal Inflammation and Perinatal Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Monica Kidd, Clinical Associate Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REB15/1418
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy

ARMS (1):
- vaccinated (Experimental): These women will have received the seasonal influenza vaccine.
  Interventions: Biological: inactivated seasonal flu vaccine

INTERVENTIONS:
Biological: inactivated seasonal flu vaccine — Women will receive the flu vaccine, and have capillary blood spots collected on day 0 and day 3.

SUMMARY:
Preventing poor perinatal outcomes is the goal of all prenatal care, yet just who will go on to develop preeclampsia or have a growth-restricted baby is notoriously difficult to predict. A growing body of evidence suggests inflammatory markers can help predict poor outcomes, even prior to, and beyond, the current pregnancy. Our project will measure the response of one robust inflammatory marker, C-reactive protein (CRP), to a safe immune provocation recommended for all pregnant women (the seasonal influenza vaccine), and to find out whether CRP response is associated with increased risk for gestational hypertension, preeclampsia, preterm delivery, or birth weight. This work will help inform whether inflammatory markers should become part of routine prenatal care.

DETAILED DESCRIPTION:
BACKGROUND

Preventing poor perinatal outcomes is the goal of all prenatal care, yet just who will go on to develop preeclampsia or have a growth-restricted baby is notoriously difficult to predict. A growing body of evidence suggests inflammatory markers can help predict poor outcomes, even prior to, and beyond, the current pregnancy. C-reactive protein (CRP) is manufactured by the liver in response to an immune provocation, and helps activate the complement system. Because it is easily assayed via phlebotomy and the less invasive capillary blood spot collection, it is a favoured marker to study inflammation in fields as diverse as immunology, obstetrics and gynecology, primary care, anthropology, and epidemiology. Pregnancy is a pro-inflammatory state, and reproductive physiology studies have shown that CRP is higher in pregnant women than in age-matched non-pregnant women, and higher still in viable pregnancies than in spontaneous abortions or ectopic pregnancies. But a look at the ecology of CRP variation shows trends with clinical relevance.

CRP is higher in obese pregnant women than in their leaner counterparts, and is positively correlated with body fat, waist-hip ratio, and HDL. While CRP does not appear to be related to insulin sensitivity in non-diabetic pregnant women, for pregnant women with type I diabetes mellitus, CRP is positively correlated with higher HgBA1C and progression of retinopathy. CRP rises with prenatal iron therapy, during labour, and during the post-partum period. It is higher for women who have had Cesarean sections than for women who delivered vaginally. And physiologic states are not the only variables associated with CRP variation. In a study of 52 women in Denver, Colorado, higher CRP was associated with higher second-trimester life stress scores and lower third-trimester social support scores. In a study of 775 women in North Carolina, higher CRP was associated with self-reported black race, qualifying for food stamps, lack of private insurance, being unmarried, previous preterm birth, and maternal weight. Does an elevated inflammatory marker also correspond to maternal or fetal morbidity?

Most research suggests it does. While one study of 32 Finnish women showed no difference in CRP between who had premature prelabour rupture of membranes (PPROM) and gestational age-matched controls, and one study of pregnant teens in New York showed CRP was associated with neither gestational age at birth nor birth weight, most studies of women in the USA, Ecuador, Colombia, the Netherlands, Hungary, Turkey, India, and South Korea have shown that higher third-trimester CRP is associated with increased risk for preeclampsia, intrauterine growth restriction, and preterm delivery. It also appears that elevated inflammatory markers may be associated with long-term maternal and infant morbidity. When CRP was tested in a prospective cohort of post-partum women who underwent diabetes screening at 3 months and 12 months post-partum, those women who developed diabetes had higher CRP at 3 months. And in Spain, high maternal CRP in the first trimester was associated with greater risk of infant wheezing and respiratory tract infections at 14 months (controlling for sex, birth weight, prematurity, maternal smoking and alcohol consumption, parity, maternal pre-pregnancy BMI, maternal total IgE, daycare attendance, and breastfeeding.

So while data on the prognostic value of CRP during pregnancy has been accumulating for more than a decade, this variable is not widely investigated in clinical obstetrics practice. Furthermore, most research has focused on static measures of CRP, not on a woman's dynamic response to an immune challenge during pregnancy because of the myriad ethical concerns with clinical trials involving pregnant women: it is possible that a woman's inflammatory response to a challenge is more clinically relevant than her baseline CRP level.

RESEARCH OBJECTIVES

The investigators propose to answer both of the above research gaps by measuring CRP response to a controlled provocation that is part of the standard of prenatal care in Canada (influenza vaccination), and to follow the results to delivery. Specifically, the investigators wish to answer the following questions:

1. What is the variation in CRP values in a cohort of pregnant women at low risk of obstetrical complications in Calgary, Alberta?
2. How does CRP respond to a standard immune provocation during pregnancy?
3. Does that response vary with age of the mother, ethnicity, gestational age, parity, BMI prior to pregnancy, and weight gain during pregnancy?
4. Does the response vary with risk of gestational hypertension, preeclampsia, preterm delivery, or birth weight?

METHODS

This will be a quantitative prospective cohort study.

Recruitment: At the beginning of 2015 flu season, the investigators will recruit participants through the low-risk prenatal clinic serving the South Health Campus in Calgary, Alberta, where the seasonal influenza vaccine is suggested as part of routine prenatal care, and where Dr. Kidd works. When women check in for their appointments, they will be given a flyer informing them of the study. Women who wish to participate in the study will be asked to present to a dedicated clinic room after their prenatal appointment, Dr. Kidd will obtain informed consent, as well as the patient's name and Alberta Health Care Number for the purpose of data retrieval. Using the standard protocol the physician will collect a capillary whole blood spot sample on Whatman #903 filter paper following a finger stick, and assign an anonymous code, e.g. 001-0. Dr. Kidd or a clinic nurse will then administer the flu vaccine. On day 3, a research assistant will obtain a second capillary blood spot sample, at the participant's home, or other convenient location. The same anonymous code will be used, e.g. 001-3. Both sets of blood spot samples, xxx-0 and xxx-3, will be sent to the Laboratory for Human Biology Research at Northwestern University, for analysis under the direction of Dr. McDade; lab personnel will not have access to participant information. Eight months later (when all participants' pregnancies will have completed), prenatal records with completed delivery information will be obtained from the electronic medical record in the clinic. Prenatal records will provide independent variables (ethnicity, gestational age, parity, BMI prior to pregnancy, and weight gain during pregnancy) and dependent variables (systolic blood pressure, diastolic blood pressure, gestational age at delivery, method of delivery, and birth weight). Any proteinuria results will be obtained through the provincial EMR, Netcare. Once datasets are complete, participants' information will be de-identified. CRP results will be added to the dataset as an additional dependent variable. The investigators will am for a convenience sample of 100 women with pre- and post-vaccination blood spots.

Laboratory analysis: The investigators will analyze blood samples for CRP (mg/L) using an improved version of a high sensitivity ELISA protocol developed specifically for dried blood spot (DBS) samples. Prior validation of assay performance indicates that the method has excellent sensitivity, precision, and reliability, and a high correlation between matched plasma and DBS samples across the entire assay range (Pearson R=0.96). For all analyses the investigators will apply standard laboratory quality control procedures, including running samples in duplicate, inspecting calibration curves for fit and day-to-day variation, and measuring quality control samples with each assay.

DATA MANAGEMENT AND ANALYSIS

All data will be kept confidential and stored in a secure location in the Department of Family Medicine at the University of Calgary. Electronic data will be password-protected. Only Dr. Kidd will have access to participant medical records, and only the research team will have access to the data.

The distribution of CRP values is likely to be skewed at baseline and day 3, and values will therefore be log transformed (base 10) to normalize the distribution. However, descriptive analyses and statistical tests will be implemented using untransformed as well as transformed results to confirm similar patterns of results. Non-parametric tests of differences in medians will be implemented using Wilcoxon matched-pairs signed-ranks and rank sum tests, and Spearman rank-order correlation will be used to assess strength of association. Log-transformed results will be subjected to paired t tests, Pearson correlation, and ordinary least squares regression analyses.

Descriptive statistics will be use to characterize baseline concentrations of CRP, and the CRP response to vaccination, in relation to prior research. Bivariate analyses will investigate the association between CRP/CRP response and the following independent variables: maternal age, ethnicity, BMI prior to pregnancy, weight gain in pregnancy, gestational age, and parity. Bivariate analyses will also investigate the association between CRP/CRP response and pregnancy complications and birth outcomes, including: systolic blood pressure, diastolic blood pressure, proteinuria, gestational age at delivery, and birth weight.

Multivariate regression analyses will investigate the associations between maternal factors and CRP/CRP response, independent of potential confounding influences. Similarly, regression analyses will investigate CRP/CRP response as independent predictors of birth outcomes.

Limitations of the study include the relatively small sample size, although prior research in this area has drawn conclusions from smaller samples. An additional limitation is the potential for loss to follow-up at two junctures: women may not be available for a research assistant to obtain a DBS on day 3, and some women's prenatal care will be transferred to obstetricians when complications arise and therefore their complete records will not be available to the research team. If it seems that too much attrition is happening before day 3, the investigators will begin asking women to collect their own DBS with disposable lancets the investigators will provide. The investigators will not be able to control for the women who are transferred to obstetrics, though Dr. Kidd's experience at the clinic is that this happens for less than 20 per cent of women initially considered to be at low-risk of complication.

ETHICAL CONSIDERATIONS

The researchers have no conflicts of interest to disclose. Health risks to participants are limited to minimal risk associated with routine vaccinations, for example pain, redness or swelling at the injection site or low-grade fever. More serious risks include allergic reaction to the vaccine (dyspnea, hives, hypotension), and Guillain-Barré syndrome, a rare ascending paralysis that affects approximately 1 in 1 million flu vaccine recipients. Risks of maternal and fetal complication from influenza are thought to far exceed risks from potential flu vaccine reaction. Risks of blood spot collection are limited to discomfort associated with a finger prick. Participants' information will be de-identified and participants will not be identified by name in any presentation or publication of study findings.

RELEVANCE

This work has important public health implications as it may help us better predict and prevent poor perinatal outcomes. For example, women with high CRP values, or high CRP responses, might benefit from closer fetal surveillance, or might need to go on medical leave earlier in their pregnancy - few guidelines are currently available to help with this clinical decision. Going forward, as new research continues to show that baseline pregnancy levels of CRP are correlated with pre-pregnancy levels, awareness of inflammatory markers in prenatal care may help us identify pre-pregnancy conditions that may lead to poor perinatal outcomes, such as social inequity and adversity. Perhaps CRP might one day be used to monitor the "readiness" of a woman contemplating pregnancy, much in the way that pre-pregnancy BMI can help predict risk of complications.

DISSEMINATION OF FINDINGS

Selected findings will be presented at appropriate venues including conferences, academic seminars and publications in the biomedical sciences and anthropology.

Our study will take place over 9 months, beginning in October, 2015.

TEAM

Dr. Monica Kidd is a family physician and low-risk obstetrics provider in Calgary, Alberta. She has a background in evolutionary biology and her research interests include child and maternal health.

Dr. Thomas McDade is a biological anthropologist specializing in human biology. His research focuses on the causes and consequences of variation in inflammation in community-based settings. He is the director of the Laboratory for Human Biology Research, which has promoted the use of dried blood spot sampling as a minimally-invasive alternative to venipuncture.

ELIGIBILITY:
Inclusion Criteria:

* Women carrying singleton pregnancies at low risk of obstetrical complication.

Exclusion Criteria:

* Pre-pregnancy BMI > 40,
* pre-existing diabetes,
* essential hypertension,
* epilepsy,
* more than one prior preterm deliveries,
* previous stillbirth,
* previous Cesarean section,
* gestational hypertension prior to 34 weeks,
* placenta previa

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-10; Primary Completion 2019-12 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
C-reactive protein (CRP) increase | three days post-vaccine compared to pre-vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Monica G Kidd, MD, Principal Investigator — (403) 956-2313
Locations (1):
- South Calgary Primary Care Network Low-Risk Maternity Clinic, Calgary, Alberta, Canada

REFERENCES:
- [Background] Breymann C, Zimmermann R, Huch R, Huch A. Use of recombinant human erythropoietin in combination with parenteral iron in the treatment of postpartum anaemia. Eur J Clin Invest. 1996 Feb;26(2):123-30. doi: 10.1046/j.1365-2362.1996.109261.x. PMID 8904521
- [Background] Christian LM, Porter K. Longitudinal changes in serum proinflammatory markers across pregnancy and postpartum: effects of maternal body mass index. Cytokine. 2014 Dec;70(2):134-40. doi: 10.1016/j.cyto.2014.06.018. Epub 2014 Jul 28. PMID 25082648
- [Background] Cicarelli LM, Perroni AG, Zugaib M, de Albuquerque PB, Campa A. Maternal and cord blood levels of serum amyloid A, C-reactive protein, tumor necrosis factor-alpha, interleukin-1beta, and interleukin-8 during and after delivery. Mediators Inflamm. 2005 Jun 9;2005(2):96-100. doi: 10.1155/MI.2005.96. PMID 16030392
- [Background] Cohen Y, Ascher-Landsberg J, Cohen A, Lessing JB, Grisaru D. The role of C-reactive protein measurement as a diagnostic aid in early pregnancy. Eur J Obstet Gynecol Reprod Biol. 2014 May;176:64-7. doi: 10.1016/j.ejogrb.2014.03.004. Epub 2014 Mar 12. PMID 24680394
- [Background] Coussons-Read ME, Okun ML, Nettles CD. Psychosocial stress increases inflammatory markers and alters cytokine production across pregnancy. Brain Behav Immun. 2007 Mar;21(3):343-50. doi: 10.1016/j.bbi.2006.08.006. Epub 2006 Oct 6. PMID 17029703
- [Background] De Meeus JB, Pourrat O, Gombert J, Magnin G. C-reactive protein levels at the onset of labour and at day 3 post-partum in normal pregnancy. Clin Exp Obstet Gynecol. 1998;25(1-2):9-11. PMID 9743869
- [Background] Derzsy Z, Prohaszka Z, Rigo J Jr, Fust G, Molvarec A. Activation of the complement system in normal pregnancy and preeclampsia. Mol Immunol. 2010 Apr;47(7-8):1500-6. doi: 10.1016/j.molimm.2010.01.021. Epub 2010 Feb 23. PMID 20181396
- [Background] Deveci K, Sogut E, Evliyaoglu O, Duras N. Pregnancy-associated plasma protein-A and C-reactive protein levels in pre-eclamptic and normotensive pregnant women at third trimester. J Obstet Gynaecol Res. 2009 Feb;35(1):94-8. doi: 10.1111/j.1447-0756.2008.00835.x. PMID 19215554
- [Background] Ernst GD, de Jonge LL, Hofman A, Lindemans J, Russcher H, Steegers EA, Jaddoe VW. C-reactive protein levels in early pregnancy, fetal growth patterns, and the risk for neonatal complications: the Generation R Study. Am J Obstet Gynecol. 2011 Aug;205(2):132.e1-12. doi: 10.1016/j.ajog.2011.03.049. Epub 2011 Apr 8. PMID 21575931
- [Background] Garcia RG, Celedon J, Sierra-Laguado J, Alarcon MA, Luengas C, Silva F, Arenas-Mantilla M, Lopez-Jaramillo P. Raised C-reactive protein and impaired flow-mediated vasodilation precede the development of preeclampsia. Am J Hypertens. 2007 Jan;20(1):98-103. doi: 10.1016/j.amjhyper.2006.06.001. PMID 17198919
- [Background] Ghosh TK, Ghosh S, Bhattacharjee D. 2011. C-reactive protein levels in women with pregnancy induced hypertension. Bangladesh Journal of Medical Science 10:159-162.
- [Background] Hwang HS, Kwon JY, Kim MA, Park YW, Kim YH. Maternal serum highly sensitive C-reactive protein in normal pregnancy and pre-eclampsia. Int J Gynaecol Obstet. 2007 Aug;98(2):105-9. doi: 10.1016/j.ijgo.2007.03.050. Epub 2007 Jun 22. PMID 17588579
- [Background] Krafft A, Perewusnyk G, Hanseler E, Quack K, Huch R, Breymann C. Effect of postpartum iron supplementation on red cell and iron parameters in non-anaemic iron-deficient women: a randomised placebo-controlled study. BJOG. 2005 Apr;112(4):445-50. doi: 10.1111/j.1471-0528.2005.00301.x. PMID 15777442
- [Background] Lohsoonthorn V, Qiu C, Williams MA. Maternal serum C-reactive protein concentrations in early pregnancy and subsequent risk of preterm delivery. Clin Biochem. 2007 Mar;40(5-6):330-5. doi: 10.1016/j.clinbiochem.2006.11.017. Epub 2007 Jan 5. PMID 17289011
- [Background] Loukovaara MJ, Alfthan HV, Kurki MT, Hiilesmaa VK, Andersson SH. Serum highly sensitive C-reactive protein in preterm premature rupture of membranes. Eur J Obstet Gynecol Reprod Biol. 2003 Sep 10;110(1):26-8. doi: 10.1016/s0301-2115(03)00084-8. PMID 12932866
- [Background] McDade TW, Williams S, Snodgrass JJ. What a drop can do: dried blood spots as a minimally invasive method for integrating biomarkers into population-based research. Demography. 2007 Nov;44(4):899-925. doi: 10.1353/dem.2007.0038. PMID 18232218
- [Background] McDade TW, Metzger MW, Chyu L, Duncan GJ, Garfield C, Adam EK. Long-term effects of birth weight and breastfeeding duration on inflammation in early adulthood. Proc Biol Sci. 2014 Apr 23;281(1784):20133116. doi: 10.1098/rspb.2013.3116. Print 2014 Jun 7. PMID 24759854
- [Background] McLachlan KA, O'Neal D, Jenkins A, Alford FP. Do adiponectin, TNFalpha, leptin and CRP relate to insulin resistance in pregnancy? Studies in women with and without gestational diabetes, during and after pregnancy. Diabetes Metab Res Rev. 2006 Mar-Apr;22(2):131-8. doi: 10.1002/dmrr.591. PMID 16170833
- [Background] Morales E, Guerra S, Garcia-Esteban R, Guxens M, Alvarez-Pedrerol M, Bustamante M, Estivill X, Anto JM, Sunyer J. Maternal C-reactive protein levels in pregnancy are associated with wheezing and lower respiratory tract infections in the offspring. Am J Obstet Gynecol. 2011 Feb;204(2):164.e1-9. doi: 10.1016/j.ajog.2010.08.056. Epub 2010 Oct 25. PMID 20974458
- [Background] Picklesimer AH, Jared HL, Moss K, Offenbacher S, Beck JD, Boggess KA. Racial differences in C-reactive protein levels during normal pregnancy. Am J Obstet Gynecol. 2008 Nov;199(5):523.e1-6. doi: 10.1016/j.ajog.2008.04.017. Epub 2008 Jun 9. PMID 18539258
- [Background] Pitiphat W, Gillman MW, Joshipura KJ, Williams PL, Douglass CW, Rich-Edwards JW. Plasma C-reactive protein in early pregnancy and preterm delivery. Am J Epidemiol. 2005 Dec 1;162(11):1108-13. doi: 10.1093/aje/kwi323. Epub 2005 Oct 19. PMID 16236995
- [Background] Ramsay JE, Ferrell WR, Crawford L, Wallace AM, Greer IA, Sattar N. Maternal obesity is associated with dysregulation of metabolic, vascular, and inflammatory pathways. J Clin Endocrinol Metab. 2002 Sep;87(9):4231-7. doi: 10.1210/jc.2002-020311. PMID 12213876
- [Background] Rebelo I, Carvalho-Guerra F, Pereira-Leite L, Quintanilha A. Lactoferrin as a sensitive blood marker of neutrophil activation in normal pregnancies. Eur J Obstet Gynecol Reprod Biol. 1995 Oct;62(2):189-94. doi: 10.1016/0301-2115(95)02203-j. PMID 8582494
- [Background] Retnakaran R, Hanley AJ, Connelly PW, Maguire G, Sermer M, Zinman B. Low serum levels of high-molecular weight adiponectin in Indo-Asian women during pregnancy: evidence of ethnic variation in adiponectin isoform distribution. Diabetes Care. 2006 Jun;29(6):1377-9. doi: 10.2337/dc06-0413. No abstract available. PMID 16732024
- [Background] Ruma M, Boggess K, Moss K, Jared H, Murtha A, Beck J, Offenbacher S. Maternal periodontal disease, systemic inflammation, and risk for preeclampsia. Am J Obstet Gynecol. 2008 Apr;198(4):389.e1-5. doi: 10.1016/j.ajog.2007.12.002. Epub 2008 Mar 4. PMID 18295179
- [Background] Spicer J, Werner E, Zhao Y, Choi CW, Lopez-Pintado S, Feng T, Altemus M, Gyamfi C, Monk C. Ambulatory assessments of psychological and peripheral stress-markers predict birth outcomes in teen pregnancy. J Psychosom Res. 2013 Oct;75(4):305-13. doi: 10.1016/j.jpsychores.2013.07.001. Epub 2013 Aug 13. PMID 24119935
- [Background] Teran E, Escudero C, Moya W, Flores M, Vallance P, Lopez-Jaramillo P. Elevated C-reactive protein and pro-inflammatory cytokines in Andean women with pre-eclampsia. Int J Gynaecol Obstet. 2001 Dec;75(3):243-9. doi: 10.1016/s0020-7292(01)00499-4. PMID 11728484
- [Background] Tjoa ML, van Vugt JM, Go AT, Blankenstein MA, Oudejans CB, van Wijk IJ. Elevated C-reactive protein levels during first trimester of pregnancy are indicative of preeclampsia and intrauterine growth restriction. J Reprod Immunol. 2003 Jun;59(1):29-37. doi: 10.1016/s0165-0378(02)00085-2. PMID 12892901
- [Background] Ustun Y, Engin-Ustun Y, Kamaci M. Association of fibrinogen and C-reactive protein with severity of preeclampsia. Eur J Obstet Gynecol Reprod Biol. 2005 Aug 1;121(2):154-8. doi: 10.1016/j.ejogrb.2004.12.009. PMID 16054955
- [Background] von Versen-Hoeynck FM, Hubel CA, Gallaher MJ, Gammill HS, Powers RW. Plasma levels of inflammatory markers neopterin, sialic acid, and C-reactive protein in pregnancy and preeclampsia. Am J Hypertens. 2009 Jun;22(6):687-92. doi: 10.1038/ajh.2009.54. Epub 2009 Mar 12. PMID 19282816
- [Background] Watts DH, Krohn MA, Wener MH, Eschenbach DA. C-reactive protein in normal pregnancy. Obstet Gynecol. 1991 Feb;77(2):176-80. doi: 10.1097/00006250-199102000-00002. PMID 1988876
- [Result] Qiu C, Luthy DA, Zhang C, Walsh SW, Leisenring WM, Williams MA. A prospective study of maternal serum C-reactive protein concentrations and risk of preeclampsia. Am J Hypertens. 2004 Feb;17(2):154-60. doi: 10.1016/j.amjhyper.2003.09.011. PMID 14751658